CLINICAL TRIAL: NCT02422849
Title: Acute Combined Care for Seniors in Southern Denmark
Acronym: ACCESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, associate professor, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SHS-ED-01-2013
Record Dates: First submitted 2015-03-27; First posted 2015-04-21 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Acute Medical Conditions
Keywords: Patient admission
MeSH Terms: interventions — General Practitioners

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- own GP (Other): The patient is cared for by own General Practitioner in the acute stage
  Interventions: Other: General Practitioner
- Hospital specialist (Other): The patient is cared for by a hospital specialist in the acute stage
  Interventions: Other: hospital specialist

INTERVENTIONS:
Other: hospital specialist
  Arms: Hospital specialist
Other: General Practitioner
  Arms: own GP

SUMMARY:
the elderly population (+ 65 years) is increasing. Acute medical conditions often leads to hospital admissions in this age group. However hospital admission is linked to adverse events. like confusion, medication errors or new infections.

the ACCESS project aims to examine alternatives to acute admissions for senior medical patients.

the aims are:

1. How many patients will be admitted to hospital due to acute medical conditions if cared for by their own General Practitioner (GP) versus a hospital intern specialist ?
2. how many patients will be admitted to hospital due to acute medical conditions if cared for by acute team in their home versus in specialised care centres ?

ELIGIBILITY:
Inclusion Criteria:

* acute medical condition requiring immediate intervention.

Exclusion Criteria:

* GP not available next days
* absolutely admission requiring condition
* no informed consent obtainable
* nursing home resident
* inclusion in ACCESS within the last 3 months
* home care capacity limit reached

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2013-11; Primary Completion 2015-02 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
number of participants with hospital admission | 3 months after inclusion

SECONDARY OUTCOMES:
change from baseline in De Morton Mobility Index (DEMMI) | 3 months after inclusion
change from baseline in quality of life (EQ5D scale) | 3 months after inclusion
change from baseline in Orientation Memory-Concentration (OMC) | 3 months after inclusion
patient and relatives satisfaction questionnaire | 3 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Aabenraa Sygehus Emergency Department, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No